CLINICAL TRIAL: NCT06265675
Title: Comparison of the Efficacy of Ultrasound-Guided Phenol Block and Corticosteroid-Local Anesthetic Block Applied to the Genicular Nerve in Patients With Knee Osteoarthritis
Brief Title: Comparison of the Efficacy of Phenol Block and Corticosteroid-Local Anesthetic Block Applied to the Genicular Nerve
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Rabia Layık, assist. dr., Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E1-4066/2023
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Genicular nerve; Phenol; Knee Osteoarthritis; Neurolysis; Nerve Blockage
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Phenol; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenol block group (Experimental)
  Interventions: Drug: Phenol
- Corticosteroid and local anesthetic (Active Comparator)
  Interventions: Drug: Celestone; Drug: Lidocain

INTERVENTIONS:
Drug: Phenol — Chemical neurolysis
  Arms: Phenol block group
Drug: Celestone — Chemical neurolysis with corticosteroid
  Arms: Corticosteroid and local anesthetic
Drug: Lidocain — Chemical neurolysis with local anesthetic
  Arms: Corticosteroid and local anesthetic

SUMMARY:
There are different neurolysis methods. Aim of this study is to compare two different methods, phenol block and corticosteroid local anesthetic block.

DETAILED DESCRIPTION:
Knee osteoarthritis is one of most frequent reason of knee pain. There are different treatment methods such as analgesic drug treatment, physical therapy techniques, intraarticular injections and neurolysis techniques. In this study, we will compare neurolysis techniques these are phenol block and corticosteroid local anesthetic block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee osteoarthritis must have pain at least 6 months
* NRS score of knee pain equal or more than 5
* At least grade 3 in Kellgren-Lawrence grading scale
* Non responsive to life style change, weight control, exercises program, medical treatment and the other conservative treatments (physical therapy, intraarticular injections)
* Decreasing at NRS score more than %50 after diagnostic block
* Those who accept the consent form

Exclusion Criteria:

* Patients who have acute knee injury
* Surgery history in knee
* Connective tissue disease that affect knee
* Sciatica
* Injection story in last 3 months
* Psychiatric or neurologic diseases that affect study
* Septic arthritis, active local or systemic infection
* Coagulopathy
* Pregnancy
* Allergic reaction

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-01-24 (Estimated); Study Completion 2025-06-24 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Before the intervention, 4 weeks after the intervention and 3 months later
  Average knee pain is assessed using an 11-point NRS with terminal descriptors of no pain (score 0) and extreme pain (score 10).

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Before the intervention, 4 weeks after the intervention and 3 months later
  We will use the WOMAC in the Likert version where question are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. So the sum of the scores ranges from 0 (the best) to 96 (the worse).
Patient Global Impression of Change (PGIC) | 4 weeks after the intervention and 3 months later
  The PGIC in pain and function will be measured with a 5-point Likert scale (1-5) on the applicable follow up visits. The patients will be asked to rate the following statements:
  Please imagine how you would have described your pain intensity before the procedure. How do you feel today as compared to baseline (Start of the study) as far as your knee pain caused by OA is concerned? Please imagine how you would have described the functionality of your knee before the procedure. How do you feel today as compared to baseline (start of the study) as far as your knee functionality caused by OA is concerned?
  The options on the Likert scale are:
  much better slightly better no change slightly worse much worse
Sixt Minute Walk Test (6MWT) | Before the intervention, 4 weeks after the intervention and 3 months later
  A 6 minute walk test is a submaximal exercise test that measures the distance walked over the span of 6 minutes.
The Timed-Up and Go test | Before the intervention, 4 weeks after the intervention and 3 months later
  This test measures the dynamic balance and functional mobility in older adults.A patient getting up from a chair from the sitting to the bipedal position, walking three meters, turning, returning, and sitting on the chair again.
Frequency of analgesic usage | Before the intervention, 4 weeks after the intervention and 3 months later
  Assessment of analgesic number that used by patient with knee osteoarthritis

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler, Ankara, Çankaya, Turkey (Türkiye)